CLINICAL TRIAL: NCT00731315
Title: Computer-Assisted Treatment in the Management of Adult Female Patients With Symptoms of Urinary Tract Infection in Emergency Departments and Community Health Centers: A Randomized Trial
Brief Title: Computer-Assisted Treatment of Urinary Tract Infection in Emergency Departments and Community Health Centers
Acronym: UTI-Kiosk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Period ended, did not reach full sample size due to limited numbers of eligible patients
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H12132-32499-02
Record Dates: First submitted 2008-08-05; First posted 2008-08-11 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Urinary Tract Infections
Keywords: UTI; Kiosk; Computer Assisted Care; cystitis
MeSH Terms: conditions — Urinary Tract Infections; Cystitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment Group 1 - uncomplicated UTI (Experimental): Would receive computer-assisted treatment for a uncomplicated UTI.
  Interventions: Other: Computer-assisted treatment group
- Control Group 1 (Active Comparator): Qualified for expedited treatment for uncomplicated cystitis but would receive usual care in the Emergency Department of Community Health Center.
  Interventions: Other: Usual care group
- Treatment Group 2 - Complicated Cystitis (Experimental): Would receive expedited treatment for complicated cystitis with longer antibiotic course than the simple UTI patients.
  Interventions: Other: Computer-assisted treatment group
- Control Group 2 (Active Comparator): Qualified for expedited treatment for complicated cystitis treatment but would receive usual care in the clinic or emergency department.
  Interventions: Other: Usual care group

INTERVENTIONS:
Other: Computer-assisted treatment group — This group will receive computer-assisted expedited treatment for uncomplicated UTI or complicated cystitis based on their symptoms and past medical history reported on the computer.
  Arms: Treatment Group 1 - uncomplicated UTI; Treatment Group 2 - Complicated Cystitis
Other: Usual care group — This group will receive usual care for an uncomplicated UTI or complicated cystitis in the Emergency Department or Community Health Center.
  Arms: Control Group 1; Control Group 2

SUMMARY:
Our study aims to test the utility of computer-assisted treatment for uncomplicated, recurrent urinary tract infections (UTIs) for women receiving care in safety net health care facilities. As of November 2009, we are also testing the utility of computer-assisted treatment for certain types of complicated cystitis (i.e. women with voiding symptoms and one of the following complicating symptoms: fever, flank pain, or symptoms greater than 7 days).

DETAILED DESCRIPTION:
An English version of the UTI Kiosk module was validated at UCSF urgent care clinic in 2005, and has been successfully integrated into the clinical work flow at this clinic for over 2 years. The computer-based module is housed in a freestanding kiosk with a touch-screen monitor and audio handset to allow patients with low literacy and minimum computer skills to complete the module. A printer in the kiosk provides a summary of the patient's responses to each question in the module, as well as a prescription for the clinic physician to sign and return to the patient.

It's important to emphasize that the computer only "fast-tracks" women who will be treated with antibiotics. All other women see the provider as usual. Also, all women who are eligible for computer treatment may opt to see a provider instead.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-64 years old

Exclusion Criteria:

* Below 18 or Above 64
* Male
* New flank pain
* severe vomiting
* High blood sugar or diabetes
* surgery on kidneys
* chronic kidney disease
* Previous cancer or chemotherapy
* HIV or AIDS
* pregnant or suspected pregnancy

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2008-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with treatment failure or relapse | 21 days

SECONDARY OUTCOMES:
Patient acceptability of treatment by computer | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Gonzales, MD, Principal Investigator — University of California, San Francsico; John Stein, MD, Principal Investigator — University of California, San Francisco; Bradley Frazee, MD, Principal Investigator — Alameda County Medical Centers, Highland Hospital
Locations (5):
- United States (5):
  - CMC Fresno Emergency Department, Fresno, California
  - La Clinica, Oakland, California
  - Highland Hospital Emergency Department, Oakland, California
  - San Francisco General Hospital - Emergency Department, San Francisco, California
  - UCSF Emergency Deparmtent, San Francisco, California